CLINICAL TRIAL: NCT00530387
Title: A Prospective, Open, Multi-Centre Photopatch Test Study of Patients Suspected of Photoallergy to Organic Sunscreens and Topical Nonsteroidal Anti-inflammatory Drugs Used Within Europe.
Brief Title: Multi-Centre European Photopatch Test Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1-Kerr
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Dermatitis, Photocontact
Keywords: Photocontact; Dermatitis; NSAID; Sunscreen; Photopatch
MeSH Terms: conditions — Dermatitis, Photoallergic; Dermatitis | interventions — homosalate; enzacamene; oxybenzone; octylmethoxycinnamate; drometrizole trisiloxane; octocrylene; 2-ethylhexyl salicylate; octyl triazone; 3-(4-methoxyphenyl)-2-propenoic acid 3-methylbutyl ester; terephthalylidene dicamphor sulfonic acid; bis-ethylhexyloxyphenol methoxyphenyl triazine; methylene bis-benzotriazolyl tetramethylphenol; diethylhexylbutamido triazone; etofenamate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 19 organic sunscreen filters and 5 topical NSAIDs
  Other Names: Butyl-methoxy-dibenzoylmethane; Homosalate; Methylbenzylidene camphor; Benzophenone-3; Octyl methoxycinnamate; Phenylbenzimidazol sulfonic acid; Benzophenone 4; Drometrizole trisiloxane; Octocrylene; Octyl salicylate; Octyl triazone; Isoamyl-p-methoxycinnamate; Terephtalidene dicamphor sulphonic acid (Mexoryl SX); Tinosorb S; Tinosorb M; Univul A+; Neoheliopan AP; Uvasorb HEB; Parsol SLX; Ketoprofen 1%; Etofenamate 2%; Piroxicam 1%; Diclofenac 5%; Ibuprofen 5 %

SUMMARY:
It is known that people can develop an allergic skin reaction to a substance which is placed on the skin and then subjected to sunlight. This process is called Photocontact allergic dermatitis. It is known that people can develop Photocontact allergic dermatitis to sunscreen chemicals (filters) and also cream forms of pain-killing drugs called nonsteroidal anti-inflammatory drugs (NSAIDs).

The purpose of this study is to determine the frequency of Photocontact allergic dermatitis to 19 sunscreen filters and 5 topical NSAIDs in 1,000 European patients who present to a dermatologist with a sun-exposed site dermatitis.

Each participant will have the 24 test agents plus one control of petrolatum applied to the skin of the back for 24 or 48 hours. After removal of the substances, the area of skin will be exposed to a precise amount of ultraviolet-A light. The area is then assessed 24, 48 and 72 hours later to see if a photocontact allergic reaction has occured. This method is known as photopatch testing.

The study will run for one year, during which time it is planned to recruit 1,000 patients.

DETAILED DESCRIPTION:
Specific Intervention Names:

* Butyl-methoxy-dibenzoylmethane
* Homosalate
* Methylbenzylidene camphor
* Benzophenone-3
* Octyl methoxycinnamate
* Phenylbenzimidazol sulfonic acid
* Benzophenone 4
* Drometrizole trisiloxane
* Octocrylene
* Octyl salicylate
* Octyl triazone
* Isoamyl-p-methoxycinnamate
* Terephtalidene dicamphor sulphonic acid (Mexoryl SX)
* Tinosorb S
* Tinosorb M
* Univul A+
* Neoheliopan AP
* Uvasorb HEB
* Parsol SLX
* Ketoprofen 1%
* Etofenamate 2%
* Piroxicam 1%
* Diclofenac 5%
* Ibuprofen 5 %

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older.
* Have sufficient cognitive capacity to give written informed consent.
* Have an eruption on photo-exposed sites, which is to be further classified using one (or more) of the categories below:
* Known photosensitivity disease
* History of sunscreen reaction
* Sun exposed site dermatitis during summer months
* Any sun exposed site dermatitis problem

Exclusion Criteria:

* Male or female aged 17 years or younger
* Have had potent topical steroid applied to the photopatch test site on the back in the previous 5 days. (This potentially suppresses reactions which would otherwise have been visible)
* Have skin disease on the back which is too active to allow testing. (This obscures the sites of testing by making differentiation between a positive result and other skin disease difficult)
* Be prescribed systemic immunosuppressant medication (e.g. prednisolone, methotrexate, azathioprine, ciclosporin) (This potentially suppresses reactions which would otherwise have been visible)
* Be taking any photoactive medicine (for example thiazides, sulphonamide derivatives, amiodarone, fluoroquinolones, chlorpromazine, NSAIDs, quinine). (This is a relative exclusion. Many centres may wish to go ahead despite such medication).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The development of a photocontact allergic skin response to sunscreen filters and topical NSAIDs, as graded by the ICDRG scale. | Within 72 hours of irradiation of patch test site

CONTACTS AND LOCATIONS:
Overall Officials: James Ferguson, FRCP, Principal Investigator — NHS Tayside
Locations (1):
- Photobiology Unit, Ninewells Hospital,, Dundee, Angus, United Kingdom